CLINICAL TRIAL: NCT06706596
Title: Implementing a Systemic Screening for TB Disease in High-risk Groups in Barcelona Area
Brief Title: A Systemic Screening for TB Disease in High-risk Groups in Barcelona
Acronym: SYS-TB-S
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Catalan Public Health Agency (Unknown); Consorci Sanitari de Barcelona (CSB) (Unknown); SMA-TB Consortium (Unknown); INNOVA4TB Consortium (Unknown); Fundació Lluita contra les Infeccions (Unknown); Hospital Vall d'Hebron -Unitat de Drassanes (Unknown); ADVANCE-TB Consortium (Unknown); Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Cris Vilaplana, Head of Tuberculosis Investigational Unit, Fundació Institut Germans Trias i Pujol
Other Study IDs: SYS-TB-S
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: Tuberculosis; Tuberculosis infection; Tuberculosis screening; Vulnerable populations; Refugees; Migrants; Pulmonary tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Latent Tuberculosis | interventions — Mass Screening; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vulnerable populations residing in the Barcelona metropolitan area with a high risk of developing TB: Individuals from vulnerable populations residing in the Barcelona metropolitan area who are at high risk of developing tuberculosis (i.e. war refugees, migrants, individuals living in socio-deprived neighborhoods)
  Interventions: Other: Screening for TB symptoms; Diagnostic Test: Chest X-ray

INTERVENTIONS:
Other: Screening for TB symptoms — Individuals will be screened for cough, blood in sputum, fever, weight loss, night sweats and chills lasting for >2 weeks
Diagnostic Test: Chest X-ray — Chest X-ray will be performed to diagnose or exclude TB

SUMMARY:
The purpose of this screening study is to identify and screen vulnerable population in Barcelona for active pulmonary tuberculosis

DETAILED DESCRIPTION:
If eligible and verbal consent is obtained, individuals:

1. Will attend a small talk/lecture about Tuberculosis (TB) disease
2. Will be interviewed and screened for the presence of TB symptoms: cough, blood in sputum, fever, weight loss, night sweats and chills lasting for >2 weeks
3. Individuals screened positive for TB will be referred to the hospital for further testing (Chest X-ray, visit, lab tests)

ELIGIBILITY:
Inclusion Criteria:

-Belonging to a population at high risk for tuberculosis (TB)

Exclusion Criteria:

-Not belonging to a population at high risk for tuberculosis (TB)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals from populations identified as high-risk for tuberculosis in the Barcelona metropolitan area
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of individuals who screen positive for pulmonary TB symptoms | 1 day
  Number of individuals who screen positive for pulmonary TB symptoms (cough, blood in sputum, fever, weight loss, night sweats and chills lasting for >2 weeks)
Number of individuals who are diagnosed with pulmonary TB symptoms | 1 month
  Number of individuals who are diagnosed with pulmonary TB symptoms after referral to the hospital

SECONDARY OUTCOMES:
Cost-effectiveness analysis | 1 day
  Cost-effectiveness analysis of the TB screening
Time spent during screening | 1 day
  Duration of each step of the screening will be analysed: duration of talk about TB, duration of waiting time before individual gets screened, duration of screening

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Vilaplana, MD, PhD, Study Chair — Fundació i Hospital Germans Trias i Pujol (IGTP-HUGTIP)
Locations (1):
- IGTP, Badalona, Spain

IPD SHARING:
Plan to Share IPD: No